CLINICAL TRIAL: NCT07368491
Title: Annual Prevalence of Airway Closure During the Full Support Phase of Invasive Mechanical Ventilation in Adults in an Intensive Care Unit
Brief Title: Prevalence of Airway Closure
Status: Not yet recruiting | Type: Observational
Sponsor: Romina Belen Mattei (Other)
Responsible Party: Sponsor-Investigator, Romina Belen Mattei, Physical Therapist, Complejo Médico Churruca Visca
Organization: Complejo Médico Churruca Visca (Other)
Other Study IDs: CEI-05092025
Record Dates: First submitted 2026-01-12; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: To Determine the Annual Prevalence of Airway Closure
Keywords: airway closure; mechanical ventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: airway closure — After setting the flow at 5 L/min and positive end-expiratory pressure (PEEP) at 0 cmH2O, the respiratory rate will be transiently decreased to achieve a prolonged expiration of 5-10 seconds to eliminate auto-PEEP. During two breaths, the change in the slope of the pressure-time curve will be observed. Airway Closure be detected as a change in the slope of the pressure-time curve. Airway Opening Pressure value, in cmH2O, will be identified on the pressure-volume curve using the cursor while the mechanical ventilator screen is frozen. Upon completion of this procedure, the ventilator settings will be returned to the patient's initial parameters.

SUMMARY:
The primary objective of this study is to describe the prevalence of airway closure during the total support phase of invasive mechanical ventilation in subjects admitted to an intensive care unit (ICU). The secondary objective is to analyze whether there are clinical-demographic and/or ventilatory characteristics associated with the presence of airway closure.

DETAILED DESCRIPTION:
Cross-sectional study. To detect airway closure, the maneuver will be performed at low flow and in case of having an opening pressure greater than 5 cmh20, the electrical impedance tomograph will be placed to record the delay in the change of impedance of each quadrant.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Requiring invasive mechanical ventilation within 48 to 72 hours after orotracheal intubation
* Hemodynamically stable (mean arterial pressure greater than 60 mmHg and/or norepinephrine less than 0.5 mcg/kg/min)
* Without respiratory muscle effort

Exclusion Criteria:

* Neumothorax
* Bronchopleural fistula
* Clinical evidence or suspicion of elevated intracranial pressure (greater than 18 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing mechanical ventilation within the first 72 hours following endotracheal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
airway closure | first 72 hours after intubation
  After setting the flow at 5 Litres/minute and positive end-expiratory pressure (PEEP) at 0 cmH2O, the respiratory rate will be transiently decreased to achieve a prolonged expiration of 5-10 seconds to eliminate auto-PEEP. During two breaths, the change in the slope of the pressure-time curve will be observed. Airway Closure be detected as a change in the slope of the pressure-time curve. Airway Opening Pressure value, in cmH2O, will be identified on the pressure-volume curve using the cursor while the mechanical ventilator screen is frozen. Upon completion of this procedure, the ventilator settings will be returned to the patient's initial parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Romina B Mattei, Principal Investigator — CMPFA Churruca-Visca
Locations (1):
- CMPFA Churruca-Visca, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided